CLINICAL TRIAL: NCT01356797
Title: Selective Unilateral Spinal Anesthesia Versus Selective Sensory Spinal Anesthesia for Knee Arthroscopy Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: USP Hospital La Colina (Other)
Responsible Party: Principal Investigator, Jesus de Santiago Moragas, MD, USP Hospital La Colina
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUAK-1
Record Dates: First submitted 2011-05-10; First posted 2011-05-19 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Pain
Keywords: knee arthroscopy; hyperbaric bupivacaine; hypobaric levobupivacaine plus fentanyl
MeSH Terms: conditions — Pain | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- hyperbaric bupivacaine (Active Comparator)
  Interventions: Drug: hyperbaric bupivacaine 0,5%
- hypobaric levobupivacaine with fentanyl (Experimental)
  Interventions: Drug: hypobaric levobupivacaine with fentanyl

INTERVENTIONS:
Drug: hypobaric levobupivacaine with fentanyl — SSSA with 4 mg hypobaric levobupivacaine 0,13% with 10 mcg fentanyl
  Other Names: Chirocane
  Arms: hypobaric levobupivacaine with fentanyl
Drug: hyperbaric bupivacaine 0,5% — SUSA with 4 mg hyperbaric bupivacaine 0.5%
  Other Names: Marchaine
  Arms: hyperbaric bupivacaine

SUMMARY:
Background: Selective unilateral spinal anesthesia is the gold standard spinal anesthesia technique for knee arthroscopy. Selective sensory spinal anesthesia has recently been validated for this surgery. Both selective techniques are specially indicated for ambulatory surgery because of PACU fast track, low discharge home time and high patient satisfaction. This study compares both spinal techniques for knee arthroscopy surgery.

ELIGIBILITY:
Inclusion Criteria:

* adults scheduled to undergo knee arthroscopy

Exclusion Criteria:

* a previous history of neurological impairment
* insulin-dependent diabetes mellitus
* intolerance to the study drug or related compounds and additives
* BMI > 38 kg/m2
* height <155 cm or >180 cm
* any existing contraindications for spinal anaesthesia
* surgery in which a complete block of the lower limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-05; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
time to discharge home | every 30 minutes for an average of 3 hours
  In Day Surgery Unit, patients will be assessed for home discharge every 30 minutes and will be followed an expected average of three hours.

SECONDARY OUTCOMES:
Ambulation time after surgery | every 30 minutes for an average of 3 hours
  In PACU and in Day Surgery Unit, patients will be assessed for unassisted ambulation every 30 minutes and will be followed an expected average of three hours.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Santiago Moragas, Principal Investigator — USP La Colina; Javier Santos-Yglesias, Study Chair — Department of Anesthesiology, Hospital La colina
Locations (1):
- Hospital La Colina, Santa Cruz de Tenerife, Santa Cruz, Spain